CLINICAL TRIAL: NCT00931970
Title: Comprehensive Prospective Study for Mode of Dialysis Therapy and Outcomes in ESRD
Brief Title: Mode of Dialysis Therapy and Outcomes in End Stage Renal Disease (ESRD)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Center for End Stage Renal Disease, Korea (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Kyungpook National University Hospital (Other); Daegu Metropolitan City, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); Medical Research Collaborating Center, Seoul, Korea (Other)
Responsible Party: Principal Investigator, Yong-Lim Kim, Professor, Clinical Research Center for End Stage Renal Disease, Korea
Other Study IDs: A-01
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: End-Stage Renal Disease
Keywords: Hemodialysis; Peritoneal dialysis; Mortality; Prospective cohort; Clinical study
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Whole blood Urine Dialysate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dialysis modality: Hemodialysis, Peritoneal dialysis

SUMMARY:
The purpose of this study is:

1. to compare complications and mortality of hemodialysis with those of peritoneal dialysis in Korean end stage renal disease (ESRD) patients; 2. to analyze the treatment effects on quality of life (QOL) by dialysis modality; and 3. to analyze cost-effectiveness by dialysis modality.

DETAILED DESCRIPTION:
The number of ESRD patients is growing at a much faster rate than the total population, with almost 1,000 (941.7) ESRD patients per one million as of 2006. The ESRD prevalence in Korea is ranked as high as 10th globally. The most common underlying diseases of ESRD in Korea include diabetes (42.3%), hypertension (16.9%), and chronic glomerulonephritis (13.0%). Diabetes and hypertension have been continuously increasing, as with a number of elderly patients due to population aging. From the examples of foreign countries with 2-to-3 fold larger dialysis population per million than Korea (ex. Japan, Taiwan, and the US), dialysis population here is forecasted to skyrocket. According to the 2003 data from the National Health Insurance Corporation that investigated diseases with high yearly treatment cost of over 5 million KRW, chronic renal failure (CRF) ranked first in both men and women. It was the single most expensive disease in 2000, with 212 billion KRW medical spending on 18,000 CRF patients, representing a significant burden to the national healthcare budget.

The ESRD Patient Registry run by the Korean Society of Nephrology (KSN) requires dialysis institutions to annually report the number of ESRD patients who receive renal replacement therapy, types of underlying disease, dialysis modality, and cause of death. Though the KSN statistics is useful as isolated epidemiological data, the program participation rate is only 60%, and cases of death are rarely reported. Clinical research on treatment or prognosis in CRF in Korea has mostly been performed by a single hospital or university, with no prospective, long-term, multi-center study performed yet.

The American Society of Nephrology, the National Kidney Foundation, and the American Association of Kidney Patients produce treatment guidelines based on effectiveness and safety proven through clinical trials. In the UK, NKRF and MRC have built databases on cardiovascular complications of chronic renal disease and outcomes with different treatment methods. Industrialized countries including the US, the UK, and Japan develop their standard treatment guidelines by thoroughly investigating etiology, progression, treatment, and cardiovascular complications and comparing effectiveness of known treatments.

The 5-year survival rate in ESRD patients in Korea is 37.8% for peritoneal dialysis patients and 65.2% for hemodialysis patients, respectively. There is a big discrepancy between patient's survival on HD and PD in Korea. However, it has been suspicious whether or not these survival data is convincing. QOL in maintenance dialysis patients is extremely low. Co-morbidity and time lost on dialysis makes it difficult to return to work while causing frequent hospitalization. Though their QOL might vary depending on country, culture, race, and dialysis modality, no multi-center study has been evaluated in Korea. CRF causes the largest per-patient health insurance reimbursement by the government, with the patient population continuously growing. Hospital stay is prolonged due to serious complications that require multi-disciplinary consultation drive up the medical cost. A cost-effectiveness study is urgently required. As in industrialized countries, the resources needed for development of the clinical practice guidelines are provided by the national government. "Effective clinical practice guidelines" will lower healthcare costs by preventing unnecessary medical practice and promote socioeconomic benefits and quality of care. The national government or related medical societies have yet to come up with a clinical practice guideline. Efforts should be made to work out "the KOREAN clinical practice guidelines" that will prevent clinical physicians from relying on foreign guidelines, which do not reflect the possibility of racial differences or was not proven to have effects on Koreans, and engaging in improper medical practices.

Our research contents are the same as below.

1. Basic data input by dialysis modality.
2. Collection of data on comorbidity and residual renal function at baseline.
3. Collection of data on referral time and history of emergent dialysis.
4. Comparative analysis of short-term QOL within 1 year of beginning dialysis.
5. Comparative analysis of complications by dialysis modality.
6. Comparative analysis of short-term patient/descriptive mortality and risk factors.
7. Creation of infection prevention and treatment guidelines in dialysis patients.
8. Comparative analysis of patient/descriptive mortality (3-year), complications, and risk factors by dialysis modality.
9. Analysis of cost-effectiveness by dialysis modality: survival rates and QOL versus cost.
10. Comparative analysis of residual renal function, its rate of decline, and survival rates by dialysis modality.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of end stage renal disease
* Must be at least 20 years of age
* Dialysis must be initiated in Korea
* Informed consent

Exclusion Criteria:

* Scheduled to receive kidney transplantation within 3 months
* Scheduled to emigrate to foreign country within 3 months
* Clinically suspected as acute renal failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident dialysis patients in Korea
Sampling Method: Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2009-07; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of all cause mortality | Within the 4 weeks after the event
  Survival
Incidence of change/termination of treatment modality | Within the 4 weeks after the event
  Incidence of change/termination dialysis modality

SECONDARY OUTCOMES:
Scores (ESKD-specific domain, physical (PCS) and mental (MCS) component summary scores) in health related quality of life mearused by the kidney disease quality of life (KDQOL)-Short Form (SF) | One year
  Scores (ESKD-specific domain, physical (PCS) and mental (MCS) component summary scores) in health related quality of life mearused by in health related quality of life mearused by the kidney disease quality of life (KDQOL)-Short Form (SF)-Each domain is rated on a scale from 0 to 100, with higher scores reflecting better HRQOL. The scores of the ESRD-targeted items are aggregated into KDCS score. The scores of the 36-Item Short Form Health Survey, a patient-reported survey of patient health, are classified into PCS score that includes items related to physical function, physical roles, pain, and general health, as well as MCS score that includes items related to emotional roles, emotional wellbeing, emotional energy, and social functioning.
Incidence of depressive symptom measured by the Beck Depression Inventory-II (BDI-II) (range: 0-63, higher scores mean worse depressive symptoms) | One year
  Incidence of depressive symptom measured by the Beck Depression Inventory-II (BDI-II) (range: 0-63, higher scores mean worse depressive symptoms)
Incidence of comorbidity measured by Charlson Comorbidity Index, Davies Comorbidity Index | One year
  Incidence of comorbidity measured by Charlson Comorbidity Index, Davies Comorbidity Index
Rate of preserved residual renal function | Six months
  Residual renal function-kt/v
Incidence of hospitalization episode and reason for hospitalization | Within the 4 weeks after the event
  Incidence of hospitalization episode and reason for hospitalization
Incidence of infection episode | Within the 4 weeks after the event
  Incidence of infection episode
Health cost | One year
  Health cost

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Lim Kim, M.D., Ph.D., Principal Investigator — Division of Nephrology and Department of Internal Medicine, Kyungpook National Univerisity Hospital, Daegu, Korea
Locations (33):
- South Korea (33):
  - Dong-A University Medical Center, Busan
  - Inje University Pusan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Wallace Memorial Baptist Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Daegu Fatima Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Daejeon St. Mary's Hospital, Daejeon
  - Holy Family Hospital, Goyang-si
  - NHIC Ilsan Hospital, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Incheon St. Mary's Hospital, Incheon
  - Cheju Halla General Hospital, Jeju City
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - National Medical Center, Seoul
  - Konkuk University, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Ehwa Womans University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - St. Paul's Hospital, Seoul
  - St. Vincent's Hospital, Suwon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Wonju Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ethier I, Hayat A, Pei J, Hawley CM, Johnson DW, Francis RS, Wong G, Craig JC, Viecelli AK, Htay H, Ng S, Leibowitz S, Cho Y. Peritoneal dialysis versus haemodialysis for people commencing dialysis. Cochrane Database Syst Rev. 2024 Jun 20;6(6):CD013800. doi: 10.1002/14651858.CD013800.pub2. PMID 38899545
- [Derived] Jung HY, Jeon Y, Kim YS, Kang SW, Yang CW, Kim NH, Noh HW, Jeon SJ, Lim JH, Choi JY, Cho JH, Park SH, Kim CD, Kim YL. Sex disparities in mortality among patients with kidney failure receiving dialysis. Sci Rep. 2022 Nov 3;12(1):18555. doi: 10.1038/s41598-022-16163-w. PMID 36329070
- [Derived] Oh HJ, Lee MJ, Lee HS, Park JT, Han SH, Yoo TH, Kim YL, Kim YS, Yang CW, Kim NH, Kang SW. NT-proBNP: is it a more significant risk factor for mortality than troponin T in incident hemodialysis patients? Medicine (Baltimore). 2014 Dec;93(27):e241. doi: 10.1097/MD.0000000000000241. PMID 25501091
- [Derived] Choi JY, Jang HM, Park J, Kim YS, Kang SW, Yang CW, Kim NH, Cho JH, Park SH, Kim CD, Kim YL; Clinical Research Center for End Stage Renal Disease (CRC for ESRD) Investigators. Survival advantage of peritoneal dialysis relative to hemodialysis in the early period of incident dialysis patients: a nationwide prospective propensity-matched study in Korea. PLoS One. 2013 Dec 30;8(12):e84257. doi: 10.1371/journal.pone.0084257. eCollection 2013. PMID 24386357